CLINICAL TRIAL: NCT00162734
Title: A Phase 3, Randomized, Open-Label Study of the Safety and Efficacy of Two Dose Levels of Interferon Alfacon-1 (Infergen, CIFN) Plus Ribavirin Administered Daily for 48 Weeks Versus No Treatment in Hepatitis C Infected Patients Who Are Nonresponders to Previous Pegylated Interferon Alfa Plus Ribavirin Therapy and During at Least 24 Weeks of No Treatment in IRHC-001
Brief Title: Daily-Dose Consensus Interferon and Ribavirin: Efficacy of Combined Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRHC-002; DIRECT 2
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic Hepatitis C; Liver; Pegylated; Interferon; Alpha; Ribavirin; Combination; Nonresponder; HCV; Infergen; SVR
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — interferon alfacon-1; Ribavirin

INTERVENTIONS:
Drug: Daily Infergen (Interferon Alfacon-1, CIFN) (9 or 15 µg) + Ribavirin (1000-1200 mg, based on body weight) PO Daily for up to 48 wks

SUMMARY:
This Phase 3 clinical study is designed to evaluate the safety, tolerability, and efficacy of two dose levels of Infergen (interferon alfacon-1, CIFN) plus Ribavirin administered daily for 48 weeks and no treatment in patients chronically infected with hepatitis C who are nonresponders to previous pegylated interferon alfa plus ribavirin therapy and participated during at least 24 weeks of no treatment in IRHC-001.

At the time of randomization into IRHC-001, the no treatment arm patients will be concurrently randomized in a 1:1 ration to receive Interferon Alfacon-1 (9 or 15 µg) + Ribavirin (both administered daily) or no treatment for up to 48 weeks. Patients will not be eligible for consideration to receive treatment in IRHC-002 until they have completed a minimum of 24 weeks of participation in IRHC-001.

The protocol and informed consent form that will be used must be approved by the Investigator's Institutional Review Board (IRB)/Independent Ethics Committee (IEC) before the study is initiated.

ELIGIBILITY:
(Abbreviated due to space constraints.)

Inclusion Criteria:

1. Signed informed consent form
2. Previously randomized to the No-Treatment Arm in IRHC-001 protocol
3. IRHC-001 no-treatment patients ho have either < 2 log10 reduction in plasma HCV RNA level by bDNA assay at Week 24 compared to baseline or detectable plasma HCV RNA by bDNA or TMA assays at Week 48
4. All patients and all potentially fertile sexual partners of patients must use 2 reliable forms of effective contraception during the study & for 6 months after cessation of the study drugs

Exclusion Criteria:

1. Patients who experienced hepatic decompensation during IRHC-001 or show laboratory, clinical, or physiologic evidence of hepatic decompensation at screening for IRHC-002
2. Patients who, in the opinion of the Investigator or the Sponsor, are not suitable candidates for enrollment or who would not comply w/the requirements of the study
3. Pregnant or lactating women
4. Male partners of women who are pregnant
5. Patients who were on any experimental protocols or therapy while participating in IRHC-001

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2005-02; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Evaluate sustained virologic response (SVR) rate of daily Infergen at two dose levels plus ribavirin and no treatment in chronically HCV-infected patients who are nonresponders to previous pegylated interferon alfa plus ribavirin therapy. | 72 weeks

SECONDARY OUTCOMES:
Evaluate safety & tolerability of therapy detailed in primary objective, and proportion of patients with (a) undetectable plasma HCV RNA levels at weeks 24 & 48 (b) abnormal baseline serum ALT levels that are normal at week 24, week 48 and weeks 48 & 72. | 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ralph T. Doyle, Study Director — Bausch Health Americas, Inc.

REFERENCES:
- See also: Daily-Dose Consensus Interferon and Ribavirin: Efficacy of Combined Therapy — http://www.directtrial.com